CLINICAL TRIAL: NCT00542555
Title: 301: A Phase 3 Study of the Analgesic Efficacy and Safety of HCT 3012: A Parallel, Randomized, Double Blind, 13 Week Placebo and Naproxen Controlled, Multicenter Study of HCT 3012 (375 mg Bid and 750 mg Bid) in Patients With Osteoarthritis of the Knee, Followed by Its Extension (301E): A Parallel, Randomized, Open-Label, Multicenter, 52-Week Follow-up Safety Study of HCT 3012 (375 mg Bid and 750 mg Bid) in Subjects With Osteoarthritis of the Knee
Brief Title: Analgesic Efficacy and Safety Study of Naproxcinod in Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NicOx (Industry)
Responsible Party: Dr Brigitte Duquesroix, Senior Director Clinical Research, NicOx
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCT3012-X-301/301E
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — naproxen-n-butyl nitrate; Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo bid (Placebo Comparator): At 13 weeks, the patients receiving placebo were re-randomized to receive either naproxcinod 375 mg bid or naproxcinod 750 mg bid in a 1:1 ratio in the 301E study.
  Interventions: Drug: Placebo
- Naproxcinod 375 mg bid (Experimental)
  Interventions: Drug: Naproxcinod 375 mg
- Naproxen 500 mg bid (Active Comparator)
  Interventions: Drug: Naproxen
- Naproxcinod 750 mg bid (Experimental)
  Interventions: Drug: Naproxcinod 750 mg

INTERVENTIONS:
Drug: Placebo — At 13 weeks, the patients receiving placebo were re-randomized to receive either naproxcinod 375 mg bid or naproxcinod 750 mg bid in a 1:1 ratio in the 301E study.
  Arms: Placebo bid
Drug: Naproxcinod 375 mg
  Arms: Naproxcinod 375 mg bid
Drug: Naproxen
  Arms: Naproxen 500 mg bid
Drug: Naproxcinod 750 mg
  Arms: Naproxcinod 750 mg bid

SUMMARY:
To study the efficacy and safety of naproxcinod vs. placebo and naproxen in the treatment of signs and symptoms of Osteoarthritis.

DETAILED DESCRIPTION:
This is a 13-week double-blind study followed by a 52-week, open-label, roll-over on active treatment study. These are randomized, parallel group, multicenter studies comparing efficacy and safety of naproxcinod, placebo and naproxen.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (40 or older) with a diagnosis of primary OA of the knee
* Must be a current chronic user of NSAIDS or acetaminophen
* Must discontinue all analgesic therapy at screening

Exclusion Criteria:

* Uncontrolled hypertension or diabetes
* Hepatic or renal impairment
* Current or expected use of anticoagulant
* A history of alcohol or drug abuse
* Candidates for imminent joint replacement
* Diagnosis of gastric or duodenal ulceration and/or history of significant gastro-duodenal bleeding, within the last 6 months
* Current medical disease that could confound or interfere with the evaluation of efficacy
* Participation within 30 days prior to screening in another investigational study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 918 (Actual)
Dates: Start 2005-12; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to show that naproxcinod is superior to placebo in relieving OA signs and symptoms in subjects with OA of the knee at 13 weeks and to collect long term safety data | 13 weeks / long term

REFERENCES:
- [Derived] Schnitzer TJ, Kivitz A, Frayssinet H, Duquesroix B. Efficacy and safety of naproxcinod in the treatment of patients with osteoarthritis of the knee: a 13-week prospective, randomized, multicenter study. Osteoarthritis Cartilage. 2010 May;18(5):629-39. doi: 10.1016/j.joca.2009.12.013. Epub 2010 Feb 16. PMID 20202489